CLINICAL TRIAL: NCT06451679
Title: An Observation Study of Postoperative Dietary Intake of Older Adult Hip Fracture Patients: a Weighed Food Diary
Brief Title: Postoperative Dietary Intake of Hip Fracture Patients
Status: Recruiting | Type: Observational
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Helen Lloyd, Principal Investigator, Teesside University
Other Study IDs: 2024 Jan 19539 LLOYD
Record Dates: First submitted 2024-06-03; First posted 2024-06-11 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Hip Fractures; Malnutrition; Comorbidities and Coexisting Conditions; Postoperative Complications
Keywords: Hip fracture; Perioperative; Surgical; Food diary; Nutrition
MeSH Terms: conditions — Hip Fractures; Malnutrition; Postoperative Complications | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — Observational prospective study

SUMMARY:
The goal of this observational study is to observe the postoperative dietary intake in older adult hip fracture patients from their day of surgery (day zero) until day three inclusive. The aims of this study are:

Primary aim:

To observe if the postoperative dietary energy intake (kJ/kcal) of older adult hip fracture patients meets Resting Energy Expenditure (REE) needs.

Secondary aims:

To explore if there is a correlation between postoperative dietary intake and length of hospital stay.

To explore the relationship between comorbidity (where reported) and postoperative dietary intake, according to dietary intake.

To explore (if) in the development of postoperative complications (infection, pressure ulcer and VTE), there is a correlation with postoperative dietary intake.

DETAILED DESCRIPTION:
A hip fracture is one of the most serious injuries that an older adult can sustain and with the current projections from the NHS Long Term Workforce plan of an increase in >85yrs by 55% and a current estimation of over 75,000 hip fractures per year in England, Northern Ireland and Wales with a 6-8% mortality rate at 1 year, this warrants further research to improve outcomes and look at methods beyond the National Hip Fracture Database (NHFD) to ascertain what more can be done to optimise and improve this patient group. Whilst ONS supplementation is used on an ad-hoc basis for patients with a high-risk malnutrition screening score of 2 using the MUST screening method, such tools can lack sensitivity and accuracy and are also not developed to identify the development of malnutrition in-hospital.

The proposed study for this protocol is an observation study of the dietary intake of older adult hip fracture patients. The study will comprise of a weighed food diary, commencing on day zero after surgery. Potential participants that will be invited will be older adult hip fracture patients (>60yrs) with a confirmed hip fracture diagnosis that requires surgical repair. The diary will consist of the researcher weighing the plate of food before and after the participant's meal as this is regarded as a more accurate measure than relying on participant recall and does not place the participant under any additional stress.

The researcher will not handle any food, and plates will be placed on a digital scale. Should a food have a specified weight - for example a yoghurt, the weight on the product will be recorded. Fluid intake will be recorded according to drinks served with meals and jugs of water per day. After each meal the researcher will weigh the plate; if it is a multiple item meal (for example meat, potatoes, and vegetables), the researcher will weigh the leftover components individually to ensure the validity of the weighed food method and to achieve the highest degree of accuracy possible. The researcher will not be present nor disrupt the participant during their meal. After their meal, the researcher will ask the participant if they have had any additional snacks and observe if they have had any assistance with their meal. Data will also be obtained regarding the times of meals, the ratio of staff to patients and if any complications have developed.

The aim of this study is to explore the postoperative dietary intake of older adult hip fracture patients until day three after surgery. This builds on research where data on hip fracture patients was taken in relation to diet, anthropometry, and biochemical indices during inpatient stays. Whilst the study was commenced in the second week post-surgery and compared against values at the week 1 admission as a baseline, the researchers observed a longer length of stay, drops in energy intake that coincided with a low BMI on admission and additionally, referrals for high-risk patients that were not actioned.

Subsequent studies have used varied interventions to explore postoperative nutrition, however a weighed food diary has yet to be used in the immediate postoperative period, which justifies the need for this study to explore nutritional intake as accurately as possible.

ELIGIBILITY:
Inclusion Criteria:

* Adults >60yrs with a confirmed diagnosis of a hip fracture requiring surgical repair.

Exclusion Criteria:

* Pathological hip fractures
* Traumatic hip fractures - such as a road traffic collision injury.
* Patients that cannot speak English due to the need for informed consent.
* Patients undergoing oncologic treatment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective older adult hip fracture patients aged 60 and over at the point of admission.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative dietary energy intake (kJ/kcal) of older adult hip fracture patients meets Resting Energy Expenditure (REE) needs. | 3 days
  REE in kJ/kcal

SECONDARY OUTCOMES:
The Correlation between comorbidity (where reported) and postoperative dietary intake, according to dietary intake. | From day of surgery until discharge from acute hospital stay, assessed up to 3 months
  Correlation between comorbidity and dietary intake
Correlation between Postoperative complications (infection, pressure ulcer and VTE), and postoperative dietary intake. | From day of surgery until discharge from acute hospital stay, assessed up to 3 months
  Link between complications and dietary intake
Postoperative dietary intake | From day of surgery until discharge from acute hospital stay, assessed up to 3 months
The length of hospital stay. | From day of surgery until discharge from acute hospital stay, assessed up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Teesside University, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No